CLINICAL TRIAL: NCT02920359
Title: Generation of Positive Biological Samples to Leuprolide Acetate for Doping Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, PhD, Parc de Salut Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMIMFTCL/LEUPRO; 2016-002719-16 (EudraCT Number)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: There Are no Conditions Under Study. Healthy Volunteers
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEUPRORELIN ACETATE (Experimental)
  Interventions: Drug: LEUPRORELIN ACETATE

INTERVENTIONS:
Drug: LEUPRORELIN ACETATE

SUMMARY:
The study consists of the generation of biological samples (in urine) positive to leuprorelin acetate for doping control by new developed methods, and establish the analytical parameters that reveal the administration of Leuprorelin acetate in healthy volunteers with these methods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged from 18 to 45 years.
2. Understanding and accepting the study procedures and signing the informed consent form.
3. A health profile devoid of organic or physiological disorders.
4. The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
5. Body mass index (BMI=weigh/height2) will range between 19 and 25 Kg/m2 and weight between 50 and 100 kg. BMI between 25 and 27 kg/m2 can be included by principal investigator criteria.

Exclusion Criteria:

1. Non compliance of the inclusion criteria.
2. History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance, similar nonapeptides or any excipients.
3. History of allergy or adverse reactions to any medication.
4. Subjects for which the drug involved in the study is counter indicated.
5. History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
6. History or clinical evidence of alcoholism, drug abuse, or regular use of psychoactive drugs.
7. Have been volunteer in another study with drugs in the last 3 months prior to start this study.
8. Have taken part in studies with blood donation in the last 2 months prior to start this study.
9. Having suffered any organic disease or major surgery in the six months prior to start this study.
10. A prior history of or presence of significant cardiovascular, neurological, haematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease that, in the investigator's opinion, considering the current state of the art, they are clinically significant, are life-threatening for the subjects and could interfere with the product assessment. Especially seizures or a history of epilepsy.
11. Regular use of any drug in the month prior to the study sessions, except for vitamins, herbal remedies or dietary supplements if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
12. Smokers of more than 20 cigarettes per day in the last 3 months prior to start this study.
13. Taking more than 40 g of alcohol per day.
14. Drinking more than 5 cups per day of coffee, tea, coke, stimulants or equivalent, or drinks containing xanthines, in the 3 months prior to start this study.
15. Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
16. Subjects with positive serology for hepatitis B, C or HIV.
17. Subjects with anormal values of testosterone or prostate-specific antigen according to age normal values.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Urine concentrations of leuprorelin acetate | From the administration to 6 hours post-administration
  Urine samples will be collected in two intervals after the administration of leuprorelin acetate (0-3h; 3-6h) in all experimental study sessions (3 consecutive days).